CLINICAL TRIAL: NCT02657551
Title: A Phase II Study Using Regorafenib as Second or Third Line Therapy in Metastatic Medullary Thyroid Cancer
Brief Title: A Study Using Regorafenib as Second or Third Line Therapy in Metastatic Medullary Thyroid Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Kartik Sehgal, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-350
Record Dates: First submitted 2015-11-09; First posted 2016-01-18 (Estimated); Results first posted 2023-11-15 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Thyroid Cancer
Keywords: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regorafenib (Experimental): Regorafenib tablets 80mg orally, once daily at predetermined dosage for 21 days per cycle
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — Regorafenib is a small molecule inhibitor of multiple membrane-bound and intracellular kinases involved in normal cellular functions and in pathologic processes.
  Other Names: Stivarga

SUMMARY:
This research study is studying a targeted therapy as a possible treatment for thyroid cancer. A targeted therapy is a type of treatment that uses drugs or other substances to identify and attack specific types of cancer cells with less harm to normal cells.

- The name of the study intervention involved in this study is regorafenib.

DETAILED DESCRIPTION:
This is a phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has approved regorafenib as a treatment for metastatic colorectal cancer and locally advanced, unresectable or metastatic gastrointestinal stromal tumor. Regorafenib has not been approved for treatment against thyroid cancer.

Regorafenib is an oral anti-tumor agent that blocks activity of a specific kind of protein involved in normal cellular functions and in pathologic processes such as tumor formation and maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.
* Age ≥ 18 years.
* Life expectancy of at least 12 weeks (3 months).
* Eastern Cooperative Oncology Group performance status of ≤1.
* Histologically or cytologically confirmed diagnosis of metastatic medullary thyroid cancer.
* Documented disease progression within 6 months prior to study registration, as defined by RECIST criteria.
* Must have at least 1 site of measurable disease by RECIST criteria, by version 1.1.
* Archival tissue block or unstained slides (from primary or metastatic site) must be available, otherwise fresh tissue biopsy sample will be collected.
* Any number of prior chemotherapies and targeted therapies are allowed.
* Patients must have received at least one prior line of targeted therapy.
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements within 3 weeks prior to study registration:

  * Total bilirubin ≤ 1.5 x the upper limits of normal (ULN)
  * Alanine aminotransferase (ALT) and aspartate amino-transferease (AST) ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer)
  * Alkaline phosphastase limit ≤ 2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer)
  * Serum creatinine ≤ 1.5 x the ULN
  * International normalized ratio (INR)/ Partial thromboplastin time (PTT) ≤ 1.5 x ULN. (Subjects who are prophylactically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists. Close monitoring of at least weekly evaluations will be performed until INR/PTT is stable based on a measurement that is pre-dose as defined by the local standard of care. (See Section 3.3)
  * Platelet count > 100000 /mm3, hemoglobin (Hb) > 9 g/dL, absolute neutrophil count (ANC) 1500/mm3. Blood transfusion to meet the inclusion criteria will not be allowed.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to study registration. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test. The definition of adequate contraception will be based on the judgment of the investigator.
* Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least 2 months after the last dose of study drug. The definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate.
* Subject must be able to swallow and retain oral medication.

Exclusion Criteria:

* Prior treatment with regorafenib.
* Previous assignment to treatment during this study. Subjects permanently withdrawn from study participation will not be allowed to re-enter study.
* Uncontrolled hypertension (systolic pressure >140 mm Hg or diastolic pressure > 90 mm Hg [NCI-CTCAE v4.0] on repeated measurement) despite optimal medical management.
* Active or clinically significant cardiac disease including:

  * Congestive heart failure - New York Heart Association (NYHA) > Class II.
  * Active coronary artery disease.
  * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin.
  * Unstable angina (anginal symptoms at rest), new-onset angina within 3 months before randomization, or myocardial infarction within 6 months before randomization.
* Evidence or history of bleeding diathesis or coagulopathy.
* Any hemorrhage or bleeding event ≥ NCI CTCAE Grade 3 within 4 weeks prior to start of study medication.
* Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) deep vein thrombosis or pulmonary embolism within 6 months of start of study treatment.
* Subjects with any previously untreated or concurrent cancer that is distinct in primary site or histology except cervical cancer in-situ, treated basal cell carcinoma, or superficial bladder tumor. Subjects surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before registration are allowed. All cancer treatments must be completed at least 3 years prior to study entry (i.e., signature date of the informed consent form).
* Patients with pheochromocytoma.
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy.
* Ongoing infection > Grade 2 NCI-CTCAE v4.0.
* Symptomatic metastatic brain or meningeal tumors.
* Presence of a non-healing wound, or non-healing ulcer, (that is not tumor related) or bone fracture.
* Major surgical procedure or significant traumatic injury within 28 days before start of study medication.
* Other investigational treatment during or within 30 days before starting study treatment.
* Use of any approved tyrosine kinase inhibitors within 2 weeks or 6 half-lives of the agen, whichever is shorter, prior to receiving study drug.
* Prior radiation within 14 days before start of study medication.Renal failure requiring hemo-or peritoneal dialysis.
* Dehydration Grade ≥1 NCI-CTCAE v4.0.
* Patients with seizure disorder requiring medication.
* Persistent proteinuria ≥ Grade 3 NCI-CTCAE v4.0 (> 3.5 g/24 hrs, measured by urine protein: creatinine ratio on a random urine sample).
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
* Pleural effusion or ascites that causes respiratory compromise (≥ NCI-CTCAE version 4.0 Grade 2 dyspnea).
* History of organ allograft (including corneal transplant).
* Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of this trial.
* Any malabsorption condition.
* Women who are pregnant or breast-feeding.
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.
* Excluded therapies and medications, previous and concomitant

  * Concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization) other than study treatment (regorafenib, other agents being investigated in combination with regorafenib).
  * Prior use of regorafenib.
  * Concurrent use of another investigational drug or device therapy (i.e., outside of study treatment) during, or within 4 weeks of trial entry (signing of the informed consent form).
  * Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study medication.
  * Therapeutic anticoagulation with Vitamin-K antagonists (e.g., warfarin) or with heparins and heparinoids.

    --- However, prophylactic anticoagulation as described below is allowed:
    * Low dose warfarin (1 mg orally, once daily) with PT-INR ≤ 1.5 x ULN is permitted. Infrequent bleeding or elevations in PT-INR have been reported in some subjects taking warfarin while on regorafenib therapy. Therefore, subjects taking concomitant warfarin should be monitored regularly for changes in PT, PT-INR or clinical bleeding episodes.
    * Low dose aspirin (≤ 100 mg daily).
    * Prophylactic doses of heparin.
  * Use of any herbal remedy (e.g. St. John's Wort [Hypericum perforatum])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Seghal, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Yale Cancer Center, New Haven, Connecticut
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data. However, at the end of the study, results will be presented and published.

REFERENCES:
- [Derived] Ettrich TJ, Seufferlein T. Regorafenib. Recent Results Cancer Res. 2018;211:45-56. doi: 10.1007/978-3-319-91442-8_3. PMID 30069758

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period: 04/21/2016-02/27/2019
Groups:
- Regorafenib Metastatic Medullary Thyroid Carcinoma (MTC): Regorafenib dose is dependent on observed significant drug related toxicities (SDRT) over cycle 1. SDRT is defined as any grade 2 or higher toxicity. For cycle 1, participants receive 80mg (2*40mg tablets) for one week. If no SDRTs, then dose is escalated to 120mg (3 tablets) for week two. Again, if no SDRTs, then dose is escalated to 160mg (4 tablets) for week three. For cycle 2-onwards, each participant received the highest tolerated dose on cycle 1. Each cycle is one daily dose for 3 weeks and 1 week off. No actual dose-escalation occurred within cycle 1 despite this potential per protocol; all participants received 80mg.
Period: Overall Study
Arm/Group | Regorafenib Metastatic Medullary Thyroid Carcinoma (MTC)
Started | 8
Completed | 0
Not Completed | 8
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Not completed — Non-Compliance | 1
Not completed — Progression / Relapse | 4

BASELINE CHARACTERISTICS:
Groups:
- Regorafenib MTC: Regorafenib dose is dependent on observed significant drug related toxicities (SDRT) over cycle 1. SDRT is defined as any grade 2 or higher toxicity. For cycle 1, participants receive 80mg (2*40mg tablets) for one week. If no SDRTs, then dose is escalated to 120mg (3 tablets) for week two. Again, if no SDRTs, then dose is escalated to 160mg (4 tablets) for week three. For cycle 2-onwards, each participant received the highest tolerated dose on cycle 1. Each cycle is one daily dose for 3 weeks and 1 week off. No actual dose-escalation occurred within cycle 1 despite this potential per protocol; all participants received 80mg.
Arm/Group | Regorafenib MTC
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (4.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4
  Asian | 1
  Other | 3
Histology [Count of Participants; unit: Participants]
  MTC | 8
  DTC | 0

OUTCOME MEASURES:

1. Primary Outcome: 10-month Progression-free Survival (PFS) Rate [MTC Cohort]
Description: 10-month PFS Rate is the proportion of participants ramaing alive and progression free at 10 months. Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) or death. Per RECIST 1.1 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease was evaluated through imaging scan on baseline, Cycle 1 Day 1, end of treatment and during follow-up. Relevant to this endpoint is 10 Months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- MTC Cohort: Regorafenib dose is dependent on observed significant drug related toxicities (SDRT) over cycle 1. SDRT is defined as any grade 2 or higher toxicity. For cycle 1, participants receive 80mg (2*40mg tablets) for one week. If no SDRTs, then dose is escalated to 120mg (3 tablets) for week two. Again, if no SDRTs, then dose is escalated to 160mg (4 tablets) for week three. For cycle 2-onwards, each participant received the highest tolerated dose on cycle 1. Each cycle is one daily dose for 3 weeks and 1 week off. No actual dose-escalation occurred within cycle 1 despite this potential per protocol; all participants received 80mg.
Arm/Group | MTC Cohort
Number analyzed (Participants) | 8
proportion of participants | 0.125 [0.003 to 0.527]

2. Primary Outcome: Response Rate [Differentiated Thyroid Cancer (DTC)] DATA NOT MATURE YET
Description: The response rate is the proportion of participants achieving XX based on RECIST 1.1 criteria defined per protocol section 11.1.4 for target lesions.
Time Frame: 2 Years
Reporting Status: Not Posted, anticipated posting 2025-12

3. Secondary Outcome: Grade 3-5 Treatment-related Toxicity Rate [MTC Cohort]
Description: All grade 3-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv4 as reported on case report forms were counted. Rate is the proportion of treated participants experiencing at least one treatment-related grade 3-5 AE of any type during the time of observation.
Time Frame: AEs were evaluated on treatment cycle 1 day 1 of week 1, 2 and 3, and cycle 2 day 1 of week 1 and 3, and cycle 3 and beyond day 1 of week 1. For this study cohort, participants were evaluated for AEs for the maximum treatment duration up to 24 months.
Measure: Number (95% Confidence Interval); unit: proportion of participant
Arm/Group | MTC Cohort
Number analyzed (Participants) | 8
proportion of participant | 0.625 [0.24 to 0.91]

4. Secondary Outcome: Quality of Life (QOL) DATA NOT MATURE YET
Description: QOL will be assessed via self-report questionnaires
Time Frame: Reported cycle 1 and 2 on day 1 of week 1 and 3, cycle 3 and beyond on day 1 of week 1, EOT, and follow-up.
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: AEs were evaluated on treatment cycle 1 day 1 of week 1, 2 and 3, and cycle 2 day 1 of week 1 and 3, and cycle 3 and beyond day 1 of week 1. For this study cohort, participants were evaluated for AEs for the maximum treatment duration of 24 months and all-cause mortality maximum follow-up of 22.5 months.
Description: Serious adverse events (AEs) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv4. All remaining events regardless of treatment attribution were classified as Other AEs. Maximum grade toxicity by type for a patient over time was calculated. No further data is available to specify classification of other beyond the general term.
Arm/Group | MTC Cohort
All-Cause Mortality (participants affected / at risk) | 4/8
Serious Adverse Events (participants affected / at risk) | 5/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MTC Cohort (N=8)
Cheilitis (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MTC Cohort (N=8)
Anemia (Blood and lymphatic system disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Dry eye (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 8
Dry mouth (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 6
Oral pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Chills (General disorders) | 1
Edema face (General disorders) | 2
Facial pain (General disorders) | 1
Fatigue (General disorders) | 5
Fever (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 5
Lymph gland infection (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Vaginal infection (Infections and infestations) | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 4
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 6
Blood bilirubin increased (Investigations) | 2
Creatinine increased (Investigations) | 2
GGT increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 2
Lymphocyte count decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Weight loss (Investigations) | 4
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 2
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 6
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT02657551/Prot_SAP_000.pdf